

Title: Drug use surveillance of Takecab tablets "Supplement to Helicobacter pylori eradication"

NCT Number: NCT03219723

Statistical analysis plan Approve Date: 08-Nov-2017

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).

Note; This document was translated into English as the language on original version was Japanese.

### Statistical Analysis Plan

(Analysis of final results)

: Supplement to *Helicobacter pylori* eradication

: Takecab Tablets

Product Name

Title of Surveillance

| Protocol No. | : Vonoprazan-5002 |
|----------------------------|-----------------------------------------|
| Sponsor | : Takeda Pharmaceutical Company Limited |
| Japan Development Center, | Takeda Pharmaceutical Company Limited |
| Head of biostatistics unit | |
| | Seal |
| Date: | |

#### Table of contents

| Li | st of | terms | s/abbreviations | 3 |
|---|---|---|---|---|
| A | nalys | is set | | 5 |
| In | nporta | ant id | entified risks, important potential risks, and important missing information | 6 |
| Н | andli | ng of | TIME WINDOW | 7 |
| Н | andli | ng of | others | 8 |
| 1 | Nur | mber | of medical institutions, number of patients enrolled, and patient disposition | 9 |
| | 1.1 | Brea | akdown of patients (figure of patient disposition) | 9 |
| 2 | Pati | ient d | emographics | 11 |
| 2 | 2.1 | Pati | ent demographics | 11 |
| 3 | Trea | atmer | nt details and concomitant drug. | 13 |
| | 3.1 | Trea | atment details | 13 |
| | 3.2 | Con | comitant drug. | 13 |
| 4 | Tab | ulate | d analysis on safety results | 14 |
| | 4.1 | Inci | dence of AE and ADR/infection | 14 |
| | 4. | .1.1 | Incidence of AE | 14 |
| | 4. | .1.2 | Incidence of ADR/infection | 14 |
| | 4. | .1.3 | Incidence of AE and ADR/infection falling under the categories of important | |
| | | | identified risks, important potential risks, and important missing information | 15 |
| | 4.2 | Inci | dence of AE and ADR/infection in patients excluded from safety evaluation | |
| | 4. | .2.1 | Incidence of AE | 17 |
| | 4. | .2.2 | Incidence of ADR/infection. | 18 |
| | 4.3 | Inci | dence of AE and ADR/infection by seriousness, time of onset, and outcome | |
| | 4. | .3.1 | Incidence of AE by seriousness, time of onset, and outcome | |
| | 4. | .3.2 | Incidence of ADR/infection by seriousness, time of onset, and outcome | 20 |
| | 4.4 | Inci | dence of ADR/infection by factor of patient demographics and treatment details | 22 |
| | 4. | .4.1 | Incidence of ADR/infection by factor of patient demographics and treatment details. | 22 |
| | 4. | .4.2 | Incidence of ADR/infection by sex | |
| | 4. | .4.3 | Incidence of ADR/infection by age subgroup | 23 |
| | 4. | .4.4 | Incidence of ADR/infection by target disease of <i>H. pylori</i> eradication | |
| | 4. | .4.5 | Incidence of ADR/infection by presence/absence of complication | |
| | 4. | .4.6 | Incidence of ADR/infection by breakdown of complication | |
| | 4. | .4.7 | Incidence of ADR/infection by BMI subgroup | |
| | 4. | .4.8 | Incidence of ADR/infection by triple therapy | |
| | | .4.9 | Incidence of ADR/infection by classification of drug | |
| | 4. | 4.10 | Incidence of ADR/infection by presence/absence of concomitant drug | 26 |

| | 4.4.11 | List of outlines of patients targeted for analysis (Attachment Form 3) | 27 |
|---|---|---|---|
| | 4.4.12 | Change of liver function test value | 28 |
| 5 | Tabulate | d analysis on efficacy results | 29 |
| | 5.1 Era | dication rate of H. pylori | 29 |
| | 5.1.1 | Eradication rate of first-line <i>H. pylori</i> eradication 4 weeks after completion of | |
| | | first-line eradication. | 29 |
| | 5.1.2 | Eradication rate of second-line <i>H. pylori</i> eradication 4 weeks after completion of | |
| | | second-line eradication | 29 |
| | 5.2 Fac | tors which may affect efficacy | 29 |
| | 5.2.1 | Eradication rate of <i>H. pylori</i> by patient demographic factor (patients of first-line | |
| | | eradication) | 29 |
| | 5.2.2 | Eradication rate of <i>H. pylori</i> by patient demographic factor (patients of second-line | |
| | | eradication) | 30 |
| Re | evision hi | story (version control) | 32 |
| ſΑ | ttachmen | t 1] Comparison Table of revision of Vonoprazan-5002 | 1 |

#### List of terms/abbreviations

- The drug: Takecab Tablets
- PPI: Proton pump inhibitor is abbreviated to PPI.
- AMPC: Amoxicillin is abbreviated to AMPC.
- CAM: Clarithromycin is abbreviated to CAM. The dose is presented as a daily dose.
- MTZ: Metronidazole is abbreviated to MTZ.
- Triple therapy: Takecab Tablets, amoxicillin and clarithromycin if it is first-line eradication. Takecab Tablets, amoxicillin and metronidazole if it is second-line eradication.
- ADR, etc.: Abbreviation of "adverse reaction and infection". Adverse events other than those
  which the surveillance investigator assessed the causality as "not related". In this statistical
  analysis plan, the term "ADR/infection" is used in the title, and the term "ADR, etc." is used in
  the text and tables.
- Serious adverse event:
  - An adverse event which the surveillance investigator assessed as "serious". Events included
    in the MedDRA code list of Takeda Medially Significant AE List are handled as serious
    even if the surveillance investigator assessed as "non-serious".
- Causality "related" to Takecab Tablets: The causality of an event assessed as "related" to Takecab Tablets or as "unassessable" is handled as "related", and the causality of an event assessed as "not related" to Takecab Tablets is handled as "not related".
- Summary statistics: An inclusive term of number of patients, mean, standard deviation, maximum value, minimum value, and quartile.
- Treatment days: The day before Takecab Tablets is started is Day -1, and the day when Takecab Tablets is started is Day 1.
- Post-treatment days: The day after the completion of Takecab Tablets administration is post-treatment Day 1.
- Patients whose survey forms have not been collected: In patients enrolled in the survey, patients whose survey forms have not been collected.
- Patients whose survey forms have been collected: In patients enrolled in this survey, patients
  whose survey forms have been collected.
- BMI (kg/m<sup>2</sup>): Calculated as Weight (kg)/Height (m)<sup>2</sup> (rounded to the first decimal place).

- Time of onset of AE (or ADR, etc.): When onset date of an AE (or ADR, etc.) is unknown, the first date of the month is the onset date. However, when the year and month of the start of Takecab Tablets and the year and month of AE (or ADR, etc.) onset are the same, the time of onset is allocated as the first start date of Takecab Tablets. The classification of time of onset is defined below when AEs (or ADRs, etc.) are counted by time of onset.
  - Duration of triple therapy: From the start day of triple therapy to the completion day of triple therapy.
  - After the completion of triple therapy: On or after the next day of the completion of triple therapy.

#### Analysis set

In this survey, two analysis sets of "safety analysis set" and "efficacy analysis set" will be set. Individual analysis sets are defined as below. Additionally, a patient enrolled and given both first-line and second-line eradication in this survey will be counted separately.

#### Safety analysis set

In this statistical analysis plan, "safety analysis set" is defined as "patients treated with Takecab Tablets with no significant protocol violation and evaluable for safety". In the patients whose survey forms have been collected, those falling under the following categories are excluded from the safety analysis set.

- Takecab Tablets was not administered
- Administration of Takecab Tablets prior to contract period
- Enrollment in this survey 6 days or later after prescription of triple therapy
- It is unknown whether any AE developed or not

#### Efficacy analysis set

In this statistical analysis plan, "efficacy analysis set" is defined as "patients treated with Takecab Tablets with no significant protocol violation and evaluable for efficacy". In the safety analysis set, patients falling under the following categories are excluded from the efficacy analysis set.

- Determination of *H. pylori* eradication has not been conducted
- Determination of *H. pylori* eradication less than 28 days after completion or discontinuation of triple therapy
- Treatment was given with a combination of three drugs other than Takecab Tablets + amoxicillin + clarithromycin in patients given first-line eradication
- Treatment was given with a combination of three drugs other than Takecab Tablets + amoxicillin + metronidazole in patients given second-line eradication

#### Important identified risks, important potential risks, and important missing information

- Important identified risk: Not applicable
- Important potential risk
  - Hepatic function disorder: An AE falling under SMQ code 20000006 (Drug related hepatic disorders - comprehensive search [SMQ] narrow) is handled as hepatic function disorder.
  - Gastrointestinal infection with clostridium difficile: An AE falling under SMQ code 20000080 (Pseudomembranous colitis [SMQ] narrow) is handled as gastrointestinal infection with clostridium difficile.
- Important missing information: Not applicable

#### **Handling of TIME WINDOW**

Data of tests/observations/endpoints which are evaluable (i.e., data which are not missing and are considered to be adopted) are handled based on the following details.

Data which are evaluable and within the time window will be adopted. If there are multiple evaluable data within the same time window, the nearest date of test/observation/assessment to the standard day will be adopted. If the number of days from the standard day is the same, data of the later date will be adopted. The difference from the standard day is determined based on the post-treatment days.

Laboratory tests (AST, ALT, γ-GTP, ALP, Total bilirubin, LDH)

| Assessment time | Standard day of conduct | Time window Post-treatment days |
|---|---|---|
| At the start of triple therapy | Post-treatment days: -1 | -8 to 1 |
| At the completion of triple therapy | Post-treatment days: 8 | 2 or more |

### Handling of others

• None particularly

#### 1 Number of medical institutions, number of patients enrolled, and patient disposition

#### 1.1 Breakdown of patients (figure of patient disposition)

Analysis All patients enrolled in this survey (patients enrolled)

population:

Analysis items: Patients enrolled

Number of medical institutions

Patients whose survey forms have not

been collected

Reason why survey form is not yet

collected

[Change of the surveillance

investigator, Health reason of the surveillance investigator, Others]

Patients whose survey forms have been

collected

Patients excluded from safety

evaluation\*

Reason of exclusion (multiple

counts)

[Takecab Tablets not administered,

Administration prior to contract period, Enrollment 6 days or later after prescription of triple therapy,

Unknown whether any AE

developed or not]

Patients targeted for safety evaluation\*

Patients excluded from efficacy

evaluation\*

Reason of exclusion (multiple

counts)

[Determination of *H. pylori* eradication

not conducted, Determination of eradication within 4 weeks after

completion or discontinuation of triple therapy, Treatment with a combination

of three drugs other than Takecab

Tablets + amoxicillin + clarithromycin in first-line eradication, Treatment with

a combination of three drugs other than

Takecab Tablets + amoxicillin + metronidazole in second-line

eradication]

Patients targeted for efficacy

evaluation\*

Analysis method: Following analysis will be conducted for the above analysis items, and a figure of patient disposition will be prepared.

> The number of medical institutions will also be calculated concerning patients enrolled in the survey. If patients are enrolled in more than one department in one medical institution, the number of the medical institution is counted as one. Number of patients excluded from safety evaluation and efficacy evaluation are counted by reason of exclusion, and a list will be prepared.

- \* "Patients targeted for safety evaluation" indicates "safety analysis set". "Patients excluded from safety evaluation" indicates patients excluded from "safety analysis set". "Patients targeted for efficacy evaluation" indicates "efficacy analysis set". "Patients excluded from efficacy evaluation" indicates patients excluded from "efficacy analysis set" in "safety analysis set".
- Frequency count

#### 2 Patient demographics

#### 2.1 Patient demographics

Analysis Safety analysis set

population:

Analysis items: Sex [Male, Female]

Age (year)  $[Min \le -.. < 65, 65 \le -.. < 75,$ 

 $75 \le - \le Max$ 

Target disease (multiple counts) [Gastric ulcer, Duodenal ulcer, Gastric

mucosa-associated lymphoid tissue
(MALT) lymphoma, Idiopathic
thrombocytopenic purpura, Stomach
following endoscopic treatment of

early gastric cancer, *H. pylori* gastritis]

Inpatient/outpatient classification [Outpatient, Inpatient]

Existence of hypersensitivity [Yes or No or Unknown]

predisposition

Existence of complication [Yes or No]

Breakdown of complication (multiple

counts) [Diabetes mellitus, Hypertension,

Lifestyle-related disease Dyslipidaemia, Hyperuricaemia]

Gastrointestinal disease (reflux

oesophagitis)

Hepatic disease [Hepatic steatosis, Alcoholic hepatitis,

Chronic hepatitis, Hepatic cirrhosis,

Viral hepatitis, Autoimmune

hepatitis]

Renal disease [Nephrotic syndrome,

Glomerulonephritis, Chronic renal

failure]

Allergic disease [Bronchial asthma, Pollinosis, Allergic

rhinitis, Allergic dermatitis]

Others

Details of previous *H. pylori* [PPI + AMPC + CAM 400 mg, PPI +

eradication AMPC + CAM 800 mg, Takecab

Tablets + AMPC + CAM 400 mg,

Takecab Tablets + AMPC + CAM 800

mg, Unknown]

Height (cm)

Weight (kg)

BMI  $(kg/m^2)$  [Min<= - <18.5, 18.5<= - <25.0,

25.0<= - <30.0, 30.0<= - <= Max ]

Smoking history [Non-smoker, Current smoker,

Ex-smoker, Unknown]

Drinking history (taking [Yes or No or Unknown]

alcohol-containing beverages almost

daily)

H. pylori infection diagnostic method

(multiple counts)

[Rapid urease test, Microscopic

method, Culture method, Urea

breath test, Anti-H. pylori antibody

assay, Stool H. pylori antigen assay]

Treatment details

First-line eradication [Takecab Tablets + AMPC + CAM,

Takecab Tablets + AMPC + MTZ]

Second-line eradication

Analysis method: Following analysis will be conducted for the above analysis items.

(1) Frequency counts of countable data, and summary statistics of quantitative data

#### 3 Treatment details and concomitant drug

#### 3.1 Treatment details

Analysis Safety analysis set

population:

Analysis items: Triple therapy [Takecab Tablets + AMPC + CAM 400]

mg, Takecab Tablets + AMPC + CAM 800 mg, Takecab Tablets + AMPC + CAM other doses, Takecab Tablets +

AMPC + MTZ

Whether triple therapy was [Yes or No]

discontinued or not

Breakdown of reasons of [Incidence of AE, No patient visit due discontinuation of triple therapy to reasons such as changing hospital,

Pregnancy, Others]

Method of determination of *H. pylori* 

eradication at the completion of triple

[Rapid urease test, Microscopic method, Culture method, Urea breath

test, Anti-H. pylori antibody assay,

Stool H. pylori antigen assay, not yet

conducted]

Analysis method: Following analysis will be conducted for the above analysis items.

(1) Frequency count

therapy (multiple counts)

#### 3.2 Concomitant drug

Analysis Safety analysis set

population:

Analysis items: Existence of concomitant drug [Yes or No]

Type of concomitant drug

Analysis method: Following analysis will be conducted for the above analysis items. Concomitant

drugs will be coded to terms in prescription drug term data file, and the data will be summarized by generic name. The drugs will be listed in descending order of frequency. When an identical drug (in generic name) is administered multiple times in one patient, one patient is counted for the drug (in generic name). When

data of a generic name is missing, the product name will be applied.

(1) Frequency count

#### 4 Tabulated analysis on safety results

#### 4.1 Incidence of AE and ADR/infection

#### 4.1.1 Incidence of AE

Analysis Safety analysis set

population:

Analysis items: Adverse event

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs
- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

• Number of patients who experienced AEs.

[Number of incidence of AEs]

 Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

#### 4.1.2 Incidence of ADR/infection

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed
multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

 To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC.
- PT will be presented with number and proportion of patients with ADRs,
   etc. in ascending order of PT codes. When multiple events coded to terms in
   an identical PT developed in a single patient, one patient will be counted for
   the PT.

# 4.1.3 Incidence of AE and ADR/infection falling under the categories of important identified risks, important potential risks, and important missing information

## 4.1.3.1 Incidence of AEs falling under the categories of important identified risks, important potential risks, and important missing information

Analysis Safety analysis set

population:

Analysis items: Adverse events falling under the categories of important identified risks,

important potential risks, and important missing information (listed in the list of

terms/abbreviations)

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs
- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

• Number of patients who experienced AEs.

[Number of incidence of AEs]

 Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

## 4.1.3.2 Incidence of ADRs/infections falling under the categories of important identified risks, important potential risks, and important missing information

Analysis Safety analysis set

population:

Analysis items: ADRs, etc. falling under the categories of important identified risks, important

potential risks, and important missing information (listed in the list of

terms/abbreviations)

Analysis method: Following analyses will be conducted for the above analysis items by drug

combination (Takecab Tablets + AMPC + CAM and Takecab Tablets + AMPC + MTZ) and pooled data of combinations.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed
multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

 To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC.
- PT will be presented with number and proportion of patients with ADRs, etc. in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

#### 4.2 Incidence of AE and ADR/infection in patients excluded from safety evaluation

#### 4.2.1 Incidence of AE

Analysis Patients excluded from safety analysis set

population:

Analysis items: Adverse event

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs

- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

• Number of patients who experienced AEs.

[Number of incidence of AEs]

• Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

#### 4.2.2 Incidence of ADR/infection

Analysis Patients excluded from safety analysis set

population:

Analysis items: ADRs, etc.

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed
multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

• To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC.
- PT will be presented with number and proportion of patients with ADRs,
   etc. in ascending order of PT codes. When multiple events coded to terms in
   an identical PT developed in a single patient, one patient will be counted for
   the PT.

#### 4.3 Incidence of AE and ADR/infection by seriousness, time of onset, and outcome

#### 4.3.1 Incidence of AE by seriousness, time of onset, and outcome

Analysis Safety analysis set

population:

Analysis items: Adverse event

Subgroup items: Seriousness [Serious, Non-serious]

Time of onset [During triple therapy, After

completion of triple therapy]

Outcome [Resolved, Resolving, Not resolved,

Resolved with sequelae, Death,

Unknown]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs
- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

• Number of patients who experienced AEs.

[Number of incidence of AEs]

• Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC. However, in an identical SOC, one event is adopted according to the priority order specified at the foot note.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT. However, for an identical PT, one event is adopted according to the following order of priority.

Seriousness: Serious → Non-serious

Time of onset: The event which developed earliest after triple therapy was started

Outcome: Death → Resolved with sequelae → Not resolved → Resolving → Resolved → Unknown

#### 4.3.2 Incidence of ADR/infection by seriousness, time of onset, and outcome

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Seriousness

tems: Seriousness [Serious, Non-serious]

Time of onset [During triple therapy, After completion of triple therapy]

20

Outcome

[Resolved, Resolving, Not resolved, Resolved with sequelae, Death, Unknown]

Analysis method: Following analyses will be conducted for the above analysis items in each subgroup by drug combination (Takecab Tablets + AMPC + CAM and Takecab Tablets + AMPC + MTZ) and pooled data of combinations.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- Proportion of patients with ADRs, etc. (3)
- **(4)** Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. ADRs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC. However, in an identical SOC, one event is adopted according to the priority order specified at the foot note.
- PT will be presented with number and proportion of patients with ADRs, etc. in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT. However, for an identical PT, one event is adopted according to the following order of priority.

Seriousness: Serious → Non-serious

Time of onset: The event which developed earliest after triple therapy was started

Outcome: Death → Resolved with sequelae → Not resolved → Resolving → Resolved → Unknown

#### 4.4 Incidence of ADR/infection by factor of patient demographics and treatment details

#### 4.4.1 Incidence of ADR/infection by factor of patient demographics and treatment details

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Sex [Male, Female]

Age (year)  $[Min \le -.. < 65, 65 \le -.. < 75,$ 

75 <= - <= Max

Target disease (multiple counts) [Gastric ulcer, Duodenal ulcer, Gastric

mucosa-associated lymphoid tissue (MALT) lymphoma, Idiopathic thrombocytopenic purpura, Stomach following endoscopic treatment of

early gastric cancer, *H. pylori* gastritis]

Existence of complication [Yes or No]

Breakdown of complication (multiple [Lifestyle-related disease,

counts) Gastrointestinal disease, Hepatic

disease, Renal disease, Allergic

disease, Others]

BMI (kg/  $m^2$ ) [Min<= - <18.5, 18.5<= - <25.0,

 $25.0 \le -30.0, 30.0 \le -8 \le Max$ 

Triple therapy [Takecab Tablets + AMPC + CAM 400

mg, Takecab Tablets + AMPC +
CAM 800 mg, Takecab Tablets +

AMPC + CAM other doses, Takecab

Tablets + AMPC + MTZ

Classification of drugs [Takecab Tablets + AMPC + CAM,

Takecab Tablets + AMPC + MTZ]

Existence of concomitant drug [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup, and chi-square test will be conducted as reference (excluding items

falling under the category of multiple counts).

(1) Number of patients with ADRs, etc.

(2) Proportion of patients with ADRs, etc. and its 95% confidence interval

(two-sided)

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Proportion of patients with ADRs, etc.]

• To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

#### 4.4.2 Incidence of ADR/infection by sex

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Sex [Male, Female]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

#### 4.4.3 Incidence of ADR/infection by age subgroup

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Age (year)  $[Min \le -.65, 65 \le -.75, \\ 75 \le -. \le Max]$ 

. .

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.4 Incidence of ADR/infection by target disease of *H. pylori* eradication

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Target disease (multiple counts) [Gastric ulcer, Duodenal ulcer, Gastric

mucosa-associated lymphoid tissue (MALT) lymphoma, Idiopathic

thrombocytopenic purpura, Stomach

following endoscopic treatment of early gastric cancer, *H. pylori* gastritis]

[Gastric ulcer or duodenal ulcer,

Gastric mucosa-associated lymphoid tissue (MALT) lymphoma or idiopathic thrombocytopenic purpura or stomach

following endoscopic treatment of early gastric cancer or *H. pylori* 

gastritis]

Analysis method: Following analyses will be conducted for the above analysis items in each

subgroup by drug combination (Takecab Tablets + AMPC + CAM and Takecab

Tablets + AMPC + MTZ) and pooled data of combinations.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.5 Incidence of ADR/infection by presence/absence of complication

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Existence of complication [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.6 Incidence of ADR/infection by breakdown of complication

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Breakdown of complication (multiple [Lifestyle-related disease,

counts) Gastrointestinal disease, Hepatic

disease, Renal disease, Allergic

disease, Others]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.7 Incidence of ADR/infection by BMI subgroup

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: BMI (kg/ m²)

 $[Min \le - <18.5, 18.5 \le - <25.0,$ 

 $25.0 \le -30.0, 30.0 \le -8 \le Max$ 

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.8 Incidence of ADR/infection by triple therapy

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Triple therapy [Takecab Tablets + AMPC + CAM 400]

mg, Takecab Tablets + AMPC + CAM 800 mg, Takecab Tablets + AMPC + CAM other doses, Takecab Tablets +

AMPC + MTZ

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

#### 4.4.9 Incidence of ADR/infection by classification of drug

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Classification of drugs [Takecab Tablets + AMPC + CAM,

Takecab Tablets + AMPC + MTZ]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

#### 4.4.10 Incidence of ADR/infection by presence/absence of concomitant drug

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Existence of concomitant drug [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

#### 4.4.11 List of outlines of patients targeted for analysis (Attachment Form 3)

Analysis Patients whose survey forms have been collected

population:

Analysis items: Patient number

Name of medical institution (company code)

Main body of establishment/code

Prefecture

Patient initials

Sex

Date of birth

Inpatient/outpatient classification

Indication (disease code, disease name)

Baseline severity

Existence of complication (yes or no, number, term)

Route of administration

Maximum dose (daily dose/one dosage)

Mean dose (daily dose/one dosage)

Unit

Daily dose frequency (maximum)

Treatment period

Concomitant drug (drug code, name of representative drug, number of drugs)

Level of effect

ADR (SOC code, ADR code, ADR term, yes or no, number)

Outcome

Survey form No.

Withdrawal

Analysis method: A list will be prepared for the above analysis items.

#### 4.4.12 Change of liver function test value

Analysis Safety analysis set

population:

Analysis items: AST (IU/L), AL T(IU/L), γ-GTP (IU/L), ALP (IU/L), Total bilirubin (mg/dL),

LDH (IU/L)

Analysis method: Summary statistics will be calculated for the measured values of each

evaluation period [at the start of triple therapy, at the completion of triple therapy] for the above analysis items. In addition, summary statistics and 95% confidence interval of mean change from the start of triple therapy will

be calculated.

#### 5 Tabulated analysis on efficacy results

#### 5.1 Eradication rate of *H. pylori*

### 5.1.1 Eradication rate of first-line *H. pylori* eradication 4 weeks after completion of first-line eradication

Analysis Patients given first-line eradication in the efficacy analysis set

population:

Analysis items: Eradication rate of first-line *H. pylori* eradication 4 weeks after completion of

first-line eradication (%)

Analysis method: Frequency will be counted for the above analysis items, and point estimates and

two-sided 95% confidence interval of eradication rates will be calculated. When

the eradication rate is calculated, the patients whose eradication is

undeterminable are excluded from the denominator.

## **5.1.2** Eradication rate of second-line *H. pylori* eradication 4 weeks after completion of second-line eradication

Analysis Patients given second-line eradication in the efficacy analysis set

population:

Analysis items: Eradication rate of second-line *H. pylori* eradication 4 weeks after the

completion of the second-line eradication (%)

Analysis method: Frequency will be counted for the above analysis items, and point estimates and

two-sided 95% confidence interval of eradication rates will be calculated. When

the eradication rate is calculated, the patients whose eradication is

undeterminable are excluded from the denominator.

#### 5.2 Factors which may affect efficacy

## 5.2.1 Eradication rate of *H. pylori* by patient demographic factor (patients of first-line eradication)

Analysis Patients given first-line eradication in the efficacy analysis set

population:

Analysis items: Eradication rate of first-line *H. pylori* eradication 4 weeks after completion of

first-line eradication (%)

Subgroup items: Sex [Male, Female]

Age (year) [Min<= - <65, 65<= - <75,

 $75 \le - \le Max$ 

Target disease (multiple counts) [Gastric ulcer, Duodenal ulcer, Gastric

mucosa-associated lymphoid tissue

(MALT) lymphoma, Idiopathic

thrombocytopenic purpura, Stomach following endoscopic treatment of early gastric cancer, *H. pylori* gastritis]

Existence of complication [Yes or No]

Breakdown of complication (multiple Lifestyle-related disease,

counts) Gastrointestinal disease, Hepatic

disease, Renal disease, Allergic

disease, Others]

BMI (kg/  $m^2$ ) [Min<= - <18.5, 18.5<= - <25.0,

25.0<= - <30.0, 30.0<= - <=Max ]

Smoking history [Non-smoker, Current smoker,

Ex-smoker, Unknown]

Drinking history (taking [Yes or No or Unknown]

alcohol-containing beverages almost

daily)

Daily dose of clarithromycin [400 mg, 800 mg, Others]

Whether triple therapy was [Yes or No]

discontinued or not

Analysis method: Frequency by each subgroup will be counted for the above analysis items, and

point estimates and two-sided 95% confidence interval of eradication rates will

be calculated. When the eradication rate is calculated, the patients whose

eradication is undeterminable are excluded from the denominator.

# 5.2.2 Eradication rate of *H. pylori* by patient demographic factor (patients of second-line eradication)

Analysis Patients given second-line eradication in the efficacy analysis set

population:

Analysis items: Eradication rate of second-line *H. pylori* eradication 4 weeks after the

completion of the second-line eradication (%)

Subgroup items: Sex [Male, Female]

Age (year) [Min<= - <65, 65<= - <75,

 $75 \le - \le Max$ 

Target disease (multiple counts) [Gastric ulcer, Duodenal ulcer, Gastric

mucosa-associated lymphoid tissue (MALT) lymphoma, Idiopathic

thrombocytopenic purpura, Stomach

following endoscopic treatment of

early gastric cancer, H. pylori gastritis]

Existence of complication [Yes or No]

Breakdown of complication (multiple [Lifestyle-related disease,

counts) Gastrointestinal disease, Hepatic

disease, Renal disease, Allergic

disease, Others]

Details of previous *H. pylori* 

eradication

[PPI + AMPC + CAM 400 mg, PPI +

AMPC + CAM 800 mg, Takecab

Tablets + AMPC + CAM 400 mg,

Takecab Tablets + AMPC + CAM 800

mg, Unknown]

BMI (kg/ $m^2$ ) [Min<= - <18.5, 18.5<= - <25.0,

25.0<= - <30.0, 30.0<= - <=Max ]

Smoking history [Non-smoker, Current smoker,

Ex-smoker, Unknown]

Drinking history (taking [Yes or No or Unknown]

alcohol-containing beverages almost

daily)

Whether triple therapy was [Yes or No]

discontinued or not

Analysis method: Frequency by each subgroup will be counted for the above analysis items, and

point estimates and two-sided 95% confidence interval of eradication rates will

be calculated. When the eradication rate is calculated, the patients whose

eradication is undeterminable are excluded from the denominator.

### **Revision history (version control)**

| Version | Date | Person who prepared/revised this document | Comment |
|---|---|---|---|
| Version 1 | August 18,<br>2017 | PPD | Preparation of Version 1 |
| Version 2 | November 8,<br>2017 | PPD | Preparation of Version 2 |

### [Attachment 1] Comparison Table of revision of Vonoprazan-5002

| Page | Before revision | After revision | Reason of revision |
|---|---|---|---|
| 10 | H. pylori infection diagnostic method (multiple counts) [Rapid urease test, Microscopic method, Culture method, Urea breath test, Anti-H. pylori antibody assay, Stool H. pylori antibody assay] | H. pylori infection diagnostic method (multiple counts) [Rapid urease test, Microscopic method, Culture method, Urea breath test, Anti-H. pylori antibody assay, Stool H. pylori antigen assay] | Correction of the incorrect term. |
| 11 | Method of determination of <i>H. pylori</i> eradication at the completion of triple therapy (multiple counts) [Rapid urease test, Microscopic method, Culture method, Urea breath test, Anti- <i>H. pylori</i> antibody assay, Stool <i>H. pylori</i> antibody assay, not yet conducted] | Method of determination of <i>H. pylori</i> eradication at the completion of triple therapy (multiple counts) [Rapid urease test, Microscopic method, Culture method, Urea breath test, Anti- <i>H. pylori</i> antibody assay, Stool <i>H. pylori</i> antigen assay, not yet conducted] | Correction of the incorrect term. |
| 11 | (New) | When data of a generic name is missing, the product name will be applied. | As there are concomitant drugs of which the drug codes are in three digits and their generic names will become missing data, it was determined to apply product names for these drugs. |

### Statistical Analysis Plan

(Analysis of final results)

: Supplement to *Helicobacter pylori* eradication

: Takecab Tablets

: Vonoprazan-5002

Product Name

Protocol No.

Title of Surveillance

| Sponsor | : Takeda Pharmaceutical Company Limited |
|----------------------------|-----------------------------------------|
| Japan Development Center, | Takeda Pharmaceutical Company Limited |
| Head of biostatistics unit | |
| | Seal |
| Date: | |
### Table of contents

| Li | st of | terms | s/abbreviations | 3 |
|---|---|---|---|---|
| A | nalys | sis set | | 5 |
| In | nporta | ant id | entified risks, important potential risks, and important missing information | 6 |
| Н | andli | ng of | TIME WINDOW | 7 |
| Н | andli | ng of | others | 8 |
| 1 | Nur | mber | of medical institutions, number of patients enrolled, and patient disposition | 9 |
| | 1.1 | Brea | akdown of patients (figure of patient disposition) | 9 |
| 2 | Pati | ient d | emographics | 11 |
| | 2.1 | Pati | ent demographics | 11 |
| 3 | Trea | atmei | nt details and concomitant drug. | 13 |
| | 3.1 | Trea | atment details | 13 |
| | 3.2 | Con | comitant drug. | 13 |
| 4 | Tab | ulate | d analysis on safety results | 14 |
| | 4.1 | Inci | dence of AE and ADR/infection | 14 |
| | 4. | .1.1 | Incidence of AE | 14 |
| | 4. | .1.2 | Incidence of ADR/infection. | 14 |
| | 4. | .1.3 | Incidence of AE and ADR/infection falling under the categories of important | |
| | | | identified risks, important potential risks, and important missing information | 15 |
| | 4.2 | Inci | dence of AE and ADR/infection in patients excluded from safety evaluation | 17 |
| | 4. | .2.1 | Incidence of AE | 17 |
| | 4. | .2.2 | Incidence of ADR/infection | 18 |
| | 4.3 | Inci | dence of AE and ADR/infection by seriousness, time of onset, and outcome | |
| | 4. | .3.1 | Incidence of AE by seriousness, time of onset, and outcome | 19 |
| | 4. | .3.2 | Incidence of ADR/infection by seriousness, time of onset, and outcome | 20 |
| | 4.4 | Inci | dence of ADR/infection by factor of patient demographics and treatment details | 22 |
| | 4. | .4.1 | Incidence of ADR/infection by factor of patient demographics and treatment details. | 22 |
| | 4. | .4.2 | Incidence of ADR/infection by sex | 23 |
| | 4. | .4.3 | Incidence of ADR/infection by age subgroup | 23 |
| | 4. | .4.4 | Incidence of ADR/infection by target disease of <i>H. pylori</i> eradication | 24 |
| | 4. | .4.5 | Incidence of ADR/infection by presence/absence of complication | 24 |
| | 4. | .4.6 | Incidence of ADR/infection by breakdown of complication | 25 |
| | 4. | .4.7 | Incidence of ADR/infection by BMI subgroup | 25 |
| | 4. | .4.8 | Incidence of ADR/infection by triple therapy | 26 |
| | | .4.9 | Incidence of ADR/infection by classification of drug | |
| | 4. | .4.10 | Incidence of ADR/infection by presence/absence of concomitant drug | 26 |

| | 4.4.11 | List of outlines of patients targeted for analysis (Attachment Form 3) | 27 |
|---|---|---|---|
| | 4.4.12 | Change of liver function test value | 28 |
| 5 Tabulated analysis on efficacy results | | | |
| | 5.1 Era | dication rate of H. pylori | 29 |
| | 5.1.1 | Eradication rate of first-line H. pylori eradication 4 weeks after completion of | |
| | | first-line eradication | 29 |
| | 5.1.2 | Eradication rate of second-line H. pylori eradication 4 weeks after completion of | |
| | | second-line eradication | 29 |
| | 5.2 Fac | tors which may affect efficacy | 29 |
| | 5.2.1 | Eradication rate of <i>H. pylori</i> by patient demographic factor (patients of first-line | |
| | | eradication) | 29 |
| | 5.2.2 | Eradication rate of <i>H. pylori</i> by patient demographic factor (patients of second-line | |
| | | eradication) | 30 |
| R | Revision history (version control) | | |
| [A | [Attachment 1] Comparison Table of revision of Vonoprazan-5002 | | |

#### List of terms/abbreviations

- The drug: Takecab Tablets
- PPI: Proton pump inhibitor is abbreviated to PPI.
- AMPC: Amoxicillin is abbreviated to AMPC.
- CAM: Clarithromycin is abbreviated to CAM. The dose is presented as a daily dose.
- MTZ: Metronidazole is abbreviated to MTZ.
- Triple therapy: Takecab Tablets, amoxicillin and clarithromycin if it is first-line eradication. Takecab Tablets, amoxicillin and metronidazole if it is second-line eradication.
- ADR, etc.: Abbreviation of "adverse reaction and infection". Adverse events other than those
  which the surveillance investigator assessed the causality as "not related". In this statistical
  analysis plan, the term "ADR/infection" is used in the title, and the term "ADR, etc." is used in
  the text and tables.
- Serious adverse event:
  - An adverse event which the surveillance investigator assessed as "serious". Events included
    in the MedDRA code list of Takeda Medially Significant AE List are handled as serious
    even if the surveillance investigator assessed as "non-serious".
- Causality "related" to Takecab Tablets: The causality of an event assessed as "related" to Takecab Tablets or as "unassessable" is handled as "related", and the causality of an event assessed as "not related" to Takecab Tablets is handled as "not related".
- Summary statistics: An inclusive term of number of patients, mean, standard deviation, maximum value, minimum value, and quartile.
- Treatment days: The day before Takecab Tablets is started is Day -1, and the day when Takecab Tablets is started is Day 1.
- Post-treatment days: The day after the completion of Takecab Tablets administration is post-treatment Day 1.
- Patients whose survey forms have not been collected: In patients enrolled in the survey, patients whose survey forms have not been collected.
- Patients whose survey forms have been collected: In patients enrolled in this survey, patients
  whose survey forms have been collected.
- BMI (kg/m<sup>2</sup>): Calculated as Weight (kg)/Height (m)<sup>2</sup> (rounded to the first decimal place).

- Time of onset of AE (or ADR, etc.): When onset date of an AE (or ADR, etc.) is unknown, the first date of the month is the onset date. However, when the year and month of the start of Takecab Tablets and the year and month of AE (or ADR, etc.) onset are the same, the time of onset is allocated as the first start date of Takecab Tablets. The classification of time of onset is defined below when AEs (or ADRs, etc.) are counted by time of onset.
  - Duration of triple therapy: From the start day of triple therapy to the completion day of triple therapy.
  - After the completion of triple therapy: On or after the next day of the completion of triple therapy.

#### Analysis set

In this survey, two analysis sets of "safety analysis set" and "efficacy analysis set" will be set. Individual analysis sets are defined as below. Additionally, a patient enrolled and given both first-line and second-line eradication in this survey will be counted separately.

#### Safety analysis set

In this statistical analysis plan, "safety analysis set" is defined as "patients treated with Takecab Tablets with no significant protocol violation and evaluable for safety". In the patients whose survey forms have been collected, those falling under the following categories are excluded from the safety analysis set.

- Takecab Tablets was not administered
- Administration of Takecab Tablets prior to contract period
- Enrollment in this survey 6 days or later after prescription of triple therapy
- It is unknown whether any AE developed or not

#### Efficacy analysis set

In this statistical analysis plan, "efficacy analysis set" is defined as "patients treated with Takecab Tablets with no significant protocol violation and evaluable for efficacy". In the safety analysis set, patients falling under the following categories are excluded from the efficacy analysis set.

- Determination of *H. pylori* eradication has not been conducted
- Determination of *H. pylori* eradication less than 28 days after completion or discontinuation of triple therapy
- Treatment was given with a combination of three drugs other than Takecab Tablets + amoxicillin + clarithromycin in patients given first-line eradication
- Treatment was given with a combination of three drugs other than Takecab Tablets + amoxicillin + metronidazole in patients given second-line eradication

#### Important identified risks, important potential risks, and important missing information

- Important identified risk: Not applicable
- Important potential risk
  - Hepatic function disorder: An AE falling under SMQ code 20000006 (Drug related hepatic disorders - comprehensive search [SMQ] narrow) is handled as hepatic function disorder.
  - Gastrointestinal infection with clostridium difficile: An AE falling under SMQ code 20000080 (Pseudomembranous colitis [SMQ] narrow) is handled as gastrointestinal infection with clostridium difficile.
- Important missing information: Not applicable

#### **Handling of TIME WINDOW**

Data of tests/observations/endpoints which are evaluable (i.e., data which are not missing and are considered to be adopted) are handled based on the following details.

Data which are evaluable and within the time window will be adopted. If there are multiple evaluable data within the same time window, the nearest date of test/observation/assessment to the standard day will be adopted. If the number of days from the standard day is the same, data of the later date will be adopted. The difference from the standard day is determined based on the post-treatment days.

Laboratory tests (AST, ALT, γ-GTP, ALP, Total bilirubin, LDH)

| Assessment time | Standard day of conduct | Time window Post-treatment days |
|---|---|---|
| At the start of triple therapy | Post-treatment days: -1 | -8 to 1 |
| At the completion of triple therapy | Post-treatment days: 8 | 2 or more |

## Handling of others

• None particularly

### 1 Number of medical institutions, number of patients enrolled, and patient disposition

#### 1.1 Breakdown of patients (figure of patient disposition)

Analysis All patients enrolled in this survey (patients enrolled)

population:

Analysis items: Patients enrolled

Number of medical institutions

Patients whose survey forms have not

been collected

Reason why survey form is not yet

collected

[Change of the surveillance

investigator, Health reason of the surveillance investigator, Others]

Patients whose survey forms have been

collected

Patients excluded from safety

evaluation\*

Reason of exclusion (multiple

counts)

[Takecab Tablets not administered,

Administration prior to contract period, Enrollment 6 days or later after prescription of triple therapy,

Unknown whether any AE

developed or not]

Patients targeted for safety evaluation\*

Patients excluded from efficacy

evaluation\*

Reason of exclusion (multiple

counts)

[Determination of *H. pylori* eradication

not conducted, Determination of eradication within 4 weeks after

completion or discontinuation of triple therapy, Treatment with a combination

of three drugs other than Takecab

Tablets + amoxicillin + clarithromycin in first-line eradication, Treatment with

a combination of three drugs other than

Takecab Tablets + amoxicillin + metronidazole in second-line

eradication]

Patients targeted for efficacy

evaluation\*

Analysis method: Following analysis will be conducted for the above analysis items, and a figure of patient disposition will be prepared.

> The number of medical institutions will also be calculated concerning patients enrolled in the survey. If patients are enrolled in more than one department in one medical institution, the number of the medical institution is counted as one. Number of patients excluded from safety evaluation and efficacy evaluation are counted by reason of exclusion, and a list will be prepared.

- \* "Patients targeted for safety evaluation" indicates "safety analysis set". "Patients excluded from safety evaluation" indicates patients excluded from "safety analysis set". "Patients targeted for efficacy evaluation" indicates "efficacy analysis set". "Patients excluded from efficacy evaluation" indicates patients excluded from "efficacy analysis set" in "safety analysis set".
- Frequency count

#### 2 Patient demographics

#### 2.1 Patient demographics

Analysis Safety analysis set

population:

Analysis items: Sex [Male, Female]

Age (year) [Min < -.. < 65, 65 < -.. < 75,

 $75 \le - \le Max$ 

Target disease (multiple counts) [Gastric ulcer, Duodenal ulcer, Gastric

mucosa-associated lymphoid tissue (MALT) lymphoma, Idiopathic

thrombocytopenic purpura, Stomach following endoscopic treatment of early gastric cancer, *H. pylori* gastritis]

Inpatient/outpatient classification [Outpatient, Inpatient]

Existence of hypersensitivity [Yes or No or Unknown]

predisposition

Existence of complication [Yes or No]

Breakdown of complication (multiple

counts)

Lifestyle-related disease [Diabetes mellitus, Hypertension,

Dyslipidaemia, Hyperuricaemia]

Gastrointestinal disease (reflux

oesophagitis)

Hepatic disease [Hepatic steatosis, Alcoholic hepatitis,

Chronic hepatitis, Hepatic cirrhosis,

Viral hepatitis, Autoimmune

hepatitis]

Renal disease [Nephrotic syndrome,

Glomerulonephritis, Chronic renal

failure]

Allergic disease [Bronchial asthma, Pollinosis, Allergic

rhinitis, Allergic dermatitis]

Others

Details of previous *H. pylori* [PPI + AMPC + CAM 400 mg, PPI +

eradication AMPC + CAM 800 mg, Takecab

Tablets + AMPC + CAM 400 mg,

Takecab Tablets + AMPC + CAM 800

mg, Unknown]

Height (cm)

Weight (kg)

BMI  $(kg/m^2)$  [Min<= - <18.5, 18.5<= - <25.0,

25.0<= - <30.0, 30.0<= - <= Max ]

Smoking history [Non-smoker, Current smoker,

Ex-smoker, Unknown]

Drinking history (taking [Yes or No or Unknown]

alcohol-containing beverages almost

daily)

H. pylori infection diagnostic method

(multiple counts)

[Rapid urease test, Microscopic method, Culture method, Urea

breath test, Anti-*H. pylori* antibody assay, Stool *H. pylori* antibody

assay]

Treatment details

First-line eradication [Takecab Tablets + AMPC + CAM,

Takecab Tablets + AMPC + MTZ]

Second-line eradication

Analysis method: Following analysis will be conducted for the above analysis items.

(1) Frequency counts of countable data, and summary statistics of quantitative data

#### 3 Treatment details and concomitant drug

#### 3.1 Treatment details

Analysis Safety analysis set

population:

Analysis items: Triple therapy [Takecab Tablets + AMPC + CAM 400]

mg, Takecab Tablets + AMPC + CAM 800 mg, Takecab Tablets + AMPC + CAM other doses, Takecab Tablets +

AMPC + MTZ

Whether triple therapy was [Yes or No]

discontinued or not

Breakdown of reasons of [Incidence of AE, No patient visit due discontinuation of triple therapy to reasons such as changing hospital,

Pregnancy, Others]

Method of determination of *H. pylori* 

eradication at the completion of triple

therapy (multiple counts) test, Anti-H. pylori antibody assay,

test, Miti-11. pytori antibody assay,

[Rapid urease test, Microscopic

method, Culture method, Urea breath

Stool *H. pylori* antibody assay, not yet

conducted]

Analysis method: Following analysis will be conducted for the above analysis items.

(1) Frequency count

#### 3.2 Concomitant drug

Analysis Safety analysis set

population:

Analysis items: Existence of concomitant drug [Yes or No]

Type of concomitant drug

Analysis method: Following analysis will be conducted for the above analysis items. Concomitant

drugs will be coded to terms in prescription drug term data file, and the data will be summarized by generic name. The drugs will be listed in descending order of frequency. When an identical drug (in generic name) is administered multiple

times in one patient, one patient is counted for the drug (in generic name).

(1) Frequency count

#### 4 Tabulated analysis on safety results

#### 4.1 Incidence of AE and ADR/infection

#### 4.1.1 Incidence of AE

Analysis Safety analysis set

population:

Analysis items: Adverse event

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs
- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

• Number of patients who experienced AEs.

[Number of incidence of AEs]

• Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

#### 4.1.2 Incidence of ADR/infection

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed
multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

 To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC.
- PT will be presented with number and proportion of patients with ADRs,
   etc. in ascending order of PT codes. When multiple events coded to terms in
   an identical PT developed in a single patient, one patient will be counted for
   the PT.

# 4.1.3 Incidence of AE and ADR/infection falling under the categories of important identified risks, important potential risks, and important missing information

# 4.1.3.1 Incidence of AEs falling under the categories of important identified risks, important potential risks, and important missing information

Analysis Safety analysis set

population:

Analysis items: Adverse events falling under the categories of important identified risks,

important potential risks, and important missing information (listed in the list of

terms/abbreviations)

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs
- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

• Number of patients who experienced AEs.

[Number of incidence of AEs]

 Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

# 4.1.3.2 Incidence of ADRs/infections falling under the categories of important identified risks, important potential risks, and important missing information

Analysis Safety analysis set

population:

Analysis items: ADRs, etc. falling under the categories of important identified risks, important

potential risks, and important missing information (listed in the list of

terms/abbreviations)

Analysis method: Following analyses will be conducted for the above analysis items by drug

combination (Takecab Tablets + AMPC + CAM and Takecab Tablets + AMPC + MTZ) and pooled data of combinations.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed
multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

 To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC.
- PT will be presented with number and proportion of patients with ADRs, etc. in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

### 4.2 Incidence of AE and ADR/infection in patients excluded from safety evaluation

#### 4.2.1 Incidence of AE

Analysis Patients excluded from safety analysis set

population:

Analysis items: Adverse event

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs

- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

• Number of patients who experienced AEs.

[Number of incidence of AEs]

• Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in
  the internationally agreed order of SOC. When multiple events coded to
  terms in an identical SOC developed in a single patient, one patient will be
  counted for the SOC.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT.

#### 4.2.2 Incidence of ADR/infection

Analysis Patients excluded from safety analysis set

population:

Analysis items: ADRs, etc.

Analysis method: Following analysis will be conducted for the above analysis items.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed
multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

• To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC.
- PT will be presented with number and proportion of patients with ADRs,
   etc. in ascending order of PT codes. When multiple events coded to terms in
   an identical PT developed in a single patient, one patient will be counted for
   the PT.

#### 4.3 Incidence of AE and ADR/infection by seriousness, time of onset, and outcome

### 4.3.1 Incidence of AE by seriousness, time of onset, and outcome

Analysis Safety analysis set

population:

Analysis items: Adverse event

Subgroup items: Seriousness [Serious, Non-serious]

Time of onset [During triple therapy, After

completion of triple therapy]

Outcome [Resolved, Resolving, Not resolved,

Resolved with sequelae, Death,

Unknown]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

- (1) Number of patients with AEs
- (2) Number of incidence of AEs
- (3) Proportion of patients with AEs
- (4) Classification of AE

The methods to count data for individual analyses are shown below.

[Number of patients with AEs]

• Number of patients who experienced AEs.

[Number of incidence of AEs]

• Number of AEs which developed. When an AE developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with AEs]

• To be calculated with number of patients with AEs/number of patients targeted for safety evaluation x 100.

[Classification of AE]

- AEs will be coded to MedDRA/J terms. AEs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with AEs in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC. However, in an identical SOC, one event is adopted according to the priority order specified at the foot note.
- PT will be presented with number and proportion of patients with AEs in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT. However, for an identical PT, one event is adopted according to the following order of priority.

Seriousness: Serious → Non-serious

Time of onset: The event which developed earliest after triple therapy was started

Outcome: Death → Resolved with sequelae → Not resolved → Resolving → Resolved → Unknown

#### 4.3.2 Incidence of ADR/infection by seriousness, time of onset, and outcome

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Seriousness [Serious, Non-serious]

Time of onset [During triple therapy, After

completion of triple therapy]

Outcome

[Resolved, Resolving, Not resolved, Resolved with sequelae, Death, Unknown]

Analysis method: Following analyses will be conducted for the above analysis items in each subgroup by drug combination (Takecab Tablets + AMPC + CAM and Takecab Tablets + AMPC + MTZ) and pooled data of combinations.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- Proportion of patients with ADRs, etc. (3)
- **(4)** Classification of ADRs, etc.

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

Number of patients who experienced ADRs, etc.

[Number of incidence of ADRs, etc.]

Number of ADRs, etc. which developed. When an ADR, etc. developed multiple times in a single patient, total number of events will be counted.

[Proportion of patients with ADRs, etc.]

To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

[Classification of ADRs, etc.]

- ADRs, etc. will be coded to MedDRA/J terms. ADRs will be counted by PT sorted by SOC. When the SOC is "Investigations", the event is counted by PT sorted by HLGT (events will be listed in ascending order of HLGT codes without output).
- SOC will be presented with number and proportion of patients with ADR, etc. in the internationally agreed order of SOC. When multiple events coded to terms in an identical SOC developed in a single patient, one patient will be counted for the SOC. However, in an identical SOC, one event is adopted according to the priority order specified at the foot note.
- PT will be presented with number and proportion of patients with ADRs, etc. in ascending order of PT codes. When multiple events coded to terms in an identical PT developed in a single patient, one patient will be counted for the PT. However, for an identical PT, one event is adopted according to the following order of priority.

Seriousness: Serious → Non-serious

Time of onset: The event which developed earliest after triple therapy was started

Outcome: Death → Resolved with sequelae → Not resolved → Resolving → Resolved → Unknown

### 4.4 Incidence of ADR/infection by factor of patient demographics and treatment details

### 4.4.1 Incidence of ADR/infection by factor of patient demographics and treatment details

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Sex [Male, Female]

Age (year) [Min<= - <65, 65<= - <75,

75 <= - <= Max

Target disease (multiple counts) [Gastric ulcer, Duodenal ulcer, Gastric

mucosa-associated lymphoid tissue (MALT) lymphoma, Idiopathic thrombocytopenic purpura, Stomach following endoscopic treatment of

early gastric cancer, *H. pylori* gastritis]

Existence of complication [Yes or No]

Breakdown of complication (multiple [Lifestyle-related disease,

counts) Gastrointestinal disease, Hepatic

disease, Renal disease, Allergic

disease, Others]

BMI (kg/  $m^2$ ) [Min<= - <18.5, 18.5<= - <25.0,

 $25.0 \le -30.0, 30.0 \le -8 \le Max$ 

Triple therapy [Takecab Tablets + AMPC + CAM 400

mg, Takecab Tablets + AMPC +
CAM 800 mg, Takecab Tablets +

AMPC + CAM other doses, Takecab

Tablets + AMPC + MTZ

Classification of drugs [Takecab Tablets + AMPC + CAM,

Takecab Tablets + AMPC + MTZ]

Existence of concomitant drug [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup, and chi-square test will be conducted as reference (excluding items

falling under the category of multiple counts).

(1) Number of patients with ADRs, etc.

(2) Proportion of patients with ADRs, etc. and its 95% confidence interval

(two-sided)

The methods to count data for individual analyses are shown below.

[Number of patients with ADRs, etc.]

• Number of patients who experienced ADRs, etc.

[Proportion of patients with ADRs, etc.]

• To be calculated with number of patients with ADRs, etc./number of patients targeted for safety evaluation x 100.

#### 4.4.2 Incidence of ADR/infection by sex

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Sex [Male, Female]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

#### 4.4.3 Incidence of ADR/infection by age subgroup

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Age (year)  $[Min \le -.. < 65, 65 \le -.. < 75,$ 

75<= - <=Max]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

#### 4.4.4 Incidence of ADR/infection by target disease of *H. pylori* eradication

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Target disease (multiple counts) [Gastric ulcer, Duodenal ulcer, Gastric

mucosa-associated lymphoid tissue (MALT) lymphoma, Idiopathic

thrombocytopenic purpura, Stomach following endoscopic treatment of

early gastric cancer, H. pylori gastritis]

[Gastric ulcer or duodenal ulcer,

Gastric mucosa-associated lymphoid tissue (MALT) lymphoma or idiopathic thrombocytopenic purpura or stomach following endoscopic treatment of early gastric cancer or *H. pylori* 

gastritis]

Analysis method: Following analyses will be conducted for the above analysis items in each subgroup by drug combination (Takecab Tablets + AMPC + CAM and Takecab

Tablets + AMPC + MTZ) and pooled data of combinations.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.
- (4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.5 Incidence of ADR/infection by presence/absence of complication

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Existence of complication [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

- (1) Number of patients with ADRs, etc.
- (2) Number of incidence of ADRs, etc.
- (3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.6 Incidence of ADR/infection by breakdown of complication

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Breakdown of complication (multiple [Lifestyle-related disease,

counts) Gastrointestinal disease, Hepatic

disease, Renal disease, Allergic

disease, Others]

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.7 Incidence of ADR/infection by BMI subgroup

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: BMI (kg/ m²)

 $[Min \le - <18.5, 18.5 \le - <25.0,]$ 

 $25.0 \le -30.0, 30.0 \le -8$ 

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in Section 4.2.2.

#### 4.4.8 Incidence of ADR/infection by triple therapy

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Triple therapy [Takecab Tablets + AMPC + CAM 400]

mg, Takecab Tablets + AMPC + CAM 800 mg, Takecab Tablets + AMPC + CAM other doses, Takecab Tablets +

AMPC + MTZ

Analysis method: Following analysis will be conducted for the above analysis items in each subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

### 4.4.9 Incidence of ADR/infection by classification of drug

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Classification of drugs [Takecab Tablets + AMPC + CAM,

Takecab Tablets + AMPC + MTZ]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

#### 4.4.10 Incidence of ADR/infection by presence/absence of concomitant drug

Analysis Safety analysis set

population:

Analysis items: ADRs, etc.

Subgroup items: Existence of concomitant drug [Yes or No]

Analysis method: Following analysis will be conducted for the above analysis items in each

subgroup.

(1) Number of patients with ADRs, etc.

(2) Number of incidence of ADRs, etc.

(3) Proportion of patients with ADRs, etc.

(4) Classification of ADRs, etc.

The methods to count individual analysis items are the same as specified in

Section 4.2.2.

#### 4.4.11 List of outlines of patients targeted for analysis (Attachment Form 3)

Analysis Patients whose survey forms have been collected

population:

Analysis items: Patient number

Name of medical institution (company code)

Main body of establishment/code

Prefecture

Patient initials

Sex

Date of birth

Inpatient/outpatient classification

Indication (disease code, disease name)

Baseline severity

Existence of complication (yes or no, number, term)

Route of administration

Maximum dose (daily dose/one dosage)

Mean dose (daily dose/one dosage)

Unit

Daily dose frequency (maximum)

Treatment period

Concomitant drug (drug code, name of representative drug, number of drugs)

Level of effect

ADR (SOC code, ADR code, ADR term, yes or no, number)

Outcome

Survey form No.

Withdrawal

Analysis method: A list will be prepared for the above analysis items.

### 4.4.12 Change of liver function test value

Analysis Safety analysis set

population:

Analysis items: AST (IU/L), AL T(IU/L), γ-GTP (IU/L), ALP (IU/L), Total bilirubin (mg/dL),

LDH (IU/L)

Analysis method: Summary statistics will be calculated for the measured values of each

evaluation period [at the start of triple therapy, at the completion of triple therapy] for the above analysis items. In addition, summary statistics and 95% confidence interval of mean change from the start of triple therapy will

be calculated.

#### 5 Tabulated analysis on efficacy results

#### 5.1 Eradication rate of *H. pylori*

# 5.1.1 Eradication rate of first-line *H. pylori* eradication 4 weeks after completion of first-line eradication

Analysis Patients given first-line eradication in the efficacy analysis set

population:

Analysis items: Eradication rate of first-line *H. pylori* eradication 4 weeks after completion of

first-line eradication (%)

Analysis method: Frequency will be counted for the above analysis items, and point estimates and

two-sided 95% confidence interval of eradication rates will be calculated. When

the eradication rate is calculated, the patients whose eradication is

undeterminable are excluded from the denominator.

# **5.1.2** Eradication rate of second-line *H. pylori* eradication 4 weeks after completion of second-line eradication

Analysis Patients given second-line eradication in the efficacy analysis set

population:

Analysis items: Eradication rate of second-line *H. pylori* eradication 4 weeks after the

completion of the second-line eradication (%)

Analysis method: Frequency will be counted for the above analysis items, and point estimates and

two-sided 95% confidence interval of eradication rates will be calculated. When

the eradication rate is calculated, the patients whose eradication is

undeterminable are excluded from the denominator.

#### 5.2 Factors which may affect efficacy

# 5.2.1 Eradication rate of *H. pylori* by patient demographic factor (patients of first-line eradication)

Analysis Patients given first-line eradication in the efficacy analysis set

population:

Analysis items: Eradication rate of first-line *H. pylori* eradication 4 weeks after completion of

first-line eradication (%)

Subgroup items: Sex [Male, Female]

Age (year) [Min<= - <65, 65<= - <75,

 $75 \le - \le Max$ 

Target disease (multiple counts) [Gastric ulcer, Duodenal ulcer, Gastric

mucosa-associated lymphoid tissue

(MALT) lymphoma, Idiopathic

thrombocytopenic purpura, Stomach following endoscopic treatment of early gastric cancer, *H. pylori* gastritis]

Existence of complication [Yes or No]

Breakdown of complication (multiple [Lifestyle-related disease,

counts) Gastrointestinal disease, Hepatic

disease, Renal disease, Allergic

disease, Others]

BMI (kg/  $m^2$ ) [Min<= - <18.5, 18.5<= - <25.0,

25.0<= - <30.0, 30.0<= - <=Max ]

Smoking history [Non-smoker, Current smoker,

Ex-smoker, Unknown]

Drinking history (taking [Yes or No or Unknown]

alcohol-containing beverages almost

daily)

Daily dose of clarithromycin [400 mg, 800 mg, Others]

Whether triple therapy was [Yes or No]

discontinued or not

Analysis method: Frequency by each subgroup will be counted for the above analysis items, and

point estimates and two-sided 95% confidence interval of eradication rates will

be calculated. When the eradication rate is calculated, the patients whose

eradication is undeterminable are excluded from the denominator.

# 5.2.2 Eradication rate of *H. pylori* by patient demographic factor (patients of second-line eradication)

Analysis Patients given second-line eradication in the efficacy analysis set

population:

Analysis items: Eradication rate of second-line *H. pylori* eradication 4 weeks after the

completion of the second-line eradication (%)

Subgroup items: Sex [Male, Female]

Age (year) [Min<= - <65, 65<= - <75,

 $75 \le - \le Max$ 

Target disease (multiple counts) [Gastric ulcer, Duodenal ulcer, Gastric

mucosa-associated lymphoid tissue (MALT) lymphoma, Idiopathic

thrombocytopenic purpura, Stomach

following endoscopic treatment of

early gastric cancer, H. pylori gastritis]

Existence of complication [Yes or No]

Breakdown of complication (multiple [Lifestyle-related disease,

counts) Gastrointestinal disease, Hepatic

disease, Renal disease, Allergic

disease, Others]

Details of previous *H. pylori* 

eradication

[PPI + AMPC + CAM 400 mg, PPI +

AMPC + CAM 800 mg, Takecab

Tablets + AMPC + CAM 400 mg,

Takecab Tablets + AMPC + CAM 800

mg, Unknown]

BMI (kg/ $m^2$ ) [Min<= -<18.5, 18.5<= -<25.0,

25.0<= - <30.0, 30.0<= - <=Max ]

Smoking history [Non-smoker, Current smoker,

Ex-smoker, Unknown]

Drinking history (taking [Yes or No or Unknown]

alcohol-containing beverages almost

daily)

Whether triple therapy was [Yes or No]

discontinued or not

Analysis method: Frequency by each subgroup will be counted for the above analysis items, and

point estimates and two-sided 95% confidence interval of eradication rates will

be calculated. When the eradication rate is calculated, the patients whose

eradication is undeterminable are excluded from the denominator.

## **Revision history (version control)**

| Version | Date | Person who prepared/revised this document | Comment |
|---|---|---|---|
| Version 1 | August 18,<br>2017 | PPD | Preparation of Version 1 |

## [Attachment 1] Comparison Table of revision of Vonoprazan-5002

Not applicable